CLINICAL TRIAL: NCT00236262
Title: Effect of the Positive Expiratory Pressure on the Right Ventricular Function in Patient With Adult Respiratory Distress Syndrome Ventilated With Limited Plateau Pressure
Brief Title: Effect of Positive Expiratory Pressure on Right Ventricular Function in Patients With Respiratory Distress Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: P040202; PS040202
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2007-03-26 (Estimated); Status verified 2007-03

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: SDRA; Distress; Expiratory; Pressure; Ventilatory
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: ventilatory strategies with pressure

SUMMARY:
The objective of this study is to analyze by trans-oesophageal echocardiography the effect on the right ventricle of positive expiratory pressure (PEP) level variations with constant plate pressure among patients with syndrome of acute respiratory distress of the adult (SDRA). The assumption tested is that a high level of PEP increases the impedance with the ejection of the right ventricle independently of the level of plate pressure. The effect on the right ventricular preload will be checked via the analysis of the respiratory variability of the diameter of the higher vena cava.

DETAILED DESCRIPTION:
Background: The ventilatory strategy in patients with Adult Respiratory Distress Syndrome (ARDS) is still controversial concerning the finest level of positive expiratory pressure (PEP). In fact, PEP allows optimisation of lung recruitment and oxygenation. However, high PEP may be detrimental on hemodynamics, notably impairing filling and ejection of the right ventricle (RV). At present, it is not known whether these adverse effects of PEP are independent or not of plateau pressure.

Objectives: The aim of the present study is to explore the effect of PEP variations (with constant plateau pressure) on RV function (assessed using trans-oesophageal echocardiography, TOE) in patients with ARDS. The assumption tested is that a high level of PEP increases the impedance to RV ejection independently of the level of plateau pressure. The effect of PEP on the right ventricular preload will also be checked via the analysis of the respiratory variability of the diameter of superior vena cava. Respiratory system properties will be assessed as follows: alveolar dead space determination using expired CO2, alveolar recruitment calculation using pressure-volume curves.

Methods: The patients are ventilated according to three consecutive strategies (A, B and C), using the same plateau pressure (<30 cm H2O), but different PEP levels: low PEP in strategy A and high PEP in strategies B and C. In order to maintain a constant plateau pressure, the increase in PEP level in strategies B and C is accompanied by a decrease in tidal volume. This decrease in tidal volume is compensated by an increase in respiratory frequency (strategy B) or a decrease of instrumental dead space by removal of heat and moisture exchanger filter (strategy C).

The first ventilatory strategy tested is "A". After that, the patient is randomised for strategies "B then C", or "C then B". At the end of each strategies the following explorations are performed: TOE, respiratory system pressure-volume curves, expired CO2 analysis, and arterial blood gas analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Intubation and artificial ventilation
2. Bilateral pulmonary opacities radiological compatible with an organic pulmonary oedema
3. PaO2/FiO2 report/ratio < 200 mmHg
4. Not obviously clinical or echocardiographic of rise in the pressure of ventricular filling left
5. Joint presence of criteria 2, 3 and 4 since less than 72 hours

Exclusion Criteria:

1. Age <18 years
2. Pregnancy
3. Obstructive chronic broncho-pneumonopathy
4. Suspected or confirmed intracranial hypertension
5. Pneumothorax
6. Evolutionary oesophageal pathology
7. Hemodynamic instability with need of filling vascular or modification of posology of the vasopressors in the 2 hours preceding inclusion
8. PaO2/FiO2 Report/ratio < 50 mmHg
9. Amount of adrenaline or noradrenaline higher than 2 mg/hour

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2005-10; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Safety
Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Laurent BROCHARD, Pr,MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- HOPITAL HENRI MONDOR Department of Neurosurgery, Créteil, France

REFERENCES:
- [Background] Bouadma L, Lellouche F, Cabello B, Taille S, Mancebo J, Dojat M, Brochard L. Computer-driven management of prolonged mechanical ventilation and weaning: a pilot study. Intensive Care Med. 2005 Oct;31(10):1446-50. doi: 10.1007/s00134-005-2766-2. Epub 2005 Aug 23. PMID 16132889
- [Background] Lacherade JC, Auburtin M, Cerf C, Van de Louw A, Soufir L, Rebufat Y, Rezaiguia S, Ricard JD, Lellouche F, Brun-Buisson C, Brochard L. Impact of humidification systems on ventilator-associated pneumonia: a randomized multicenter trial. Am J Respir Crit Care Med. 2005 Nov 15;172(10):1276-82. doi: 10.1164/rccm.200408-1028OC. Epub 2005 Aug 26. PMID 16126933
- [Derived] Mekontso Dessap A, Charron C, Devaquet J, Aboab J, Jardin F, Brochard L, Vieillard-Baron A. Impact of acute hypercapnia and augmented positive end-expiratory pressure on right ventricle function in severe acute respiratory distress syndrome. Intensive Care Med. 2009 Nov;35(11):1850-8. doi: 10.1007/s00134-009-1569-2. Epub 2009 Aug 4. PMID 19652953